CLINICAL TRIAL: NCT06539260
Title: Clinical Relationship Between Vitamin D-mediated Th17 and Treg Cells and Parkinson's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Suzhou Municipal Hospital of Anhui Province (Other)
Responsible Party: Principal Investigator, Xibo Ma, learned scholar, Suzhou Municipal Hospital of Anhui Province
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SuzhouAnhuiPD; AHWJ2022b106 (Other: Anhui Provincial Health Commission)
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Neurology; Immunology
Keywords: Parkinson's disease; Vitamin D; Treg; Th17
MeSH Terms: conditions — Parkinson Disease | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VitD group (Experimental): The Parkinson's disease patients included in the study underwent analysis of peripheral blood vitamin D levels, among other assessments. Patients with low vitamin D levels (Vit D < 30 ng/ml) were randomly assigned in a 1:1 ratio to two groups: one receiving vitamin D3 and the other receiving a placebo (PL). The vitamin D group was supplemented with vitamin D for a period of 3 months.
  Interventions: Drug: Vitamin D
- PL group (Placebo Comparator): The Parkinson's disease patients included in the study underwent analysis of peripheral blood vitamin D levels, among other assessments. Patients with low vitamin D levels (Vit D < 30 ng/ml) were randomly assigned in a 1:1 ratio to two groups: one receiving vitamin D3 and the other receiving a placebo (PL). The placebo group was supplemented with a placebo for a period of 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — Take 400 units of vitamin D3, twice daily, for a duration of 3 months.
  Arms: VitD group
Drug: Placebo — Take a placebo that is identical in appearance and weight to 400 units of vitamin D3, twice daily, for a duration of 3 months.
  Arms: PL group

SUMMARY:
The aim of this study is to detect the expression levels of vitamin D, Treg, and Th17 in the peripheral blood of patients with Parkinson's disease (PD), investigate the impact of Treg/Th17 imbalance on PD patients, and explore the effects of vitamin D intervention on Treg/Th17 imbalance and clinical outcomes. Furthermore, this study aims to delve into the potential mechanisms of vitamin D deficiency and Treg/Th17 imbalance in the pathogenesis of Parkinson's disease, ultimately providing new theoretical evidence for the research, prevention, and treatment of PD.

DETAILED DESCRIPTION:
FromJanuary 2023 to July 2024, 50 PD patients and 50 health control groups were collected. All subjects were from the Parkinson's outpatient clinic and ward of the Department of Neurology, Suzhou Hospital Affiliated to Anhui Medical University. This study was approved by the Medical Ethics Committee of Suzhou Municipal Hospital and signed an informed consent form. The gender, age, identity registration, place of origin, marital status, education level, occupation, smoking, drinking, occupational exposure, body mass index, home address and contact information of the patients were collected for detailed registration. Current medical history, past history, family history, medication use, physical examination, previous relevant auxiliary examination results, etc. Evaluation scales: H-Y Staging Scale, UPDRS Scale, Breg Balance Scale, MMSE Intelligence Scale, MoCA Scale, SDS Depression Self-Rating Scale, SAS Anxiety Self-Rating Scale, PDSS Parkinson's Disease Sleep Scale. Peripheral blood of patients and control groups were sampled to determine the levels of vitamin D, Treg and Th17. PD patients were divided into vitamin D deficiency group and vitamin D non-deficiency group according to the detection of vitamin D. Vitamin D deficiency group was randomly divided into intervention group and non-intervention group. The intervention group was supplemented with vitamin D, and the non-intervention group was not treated. The above scale and peripheral blood vitamin D, Treg and Th17 levels were evaluated after 3 months of follow-up and compared with the pre-intervention and non-intervention groups. Statistical analysis was carried out using SPSS26.0 and GraphPad Prism v.9.

ELIGIBILITY:
Inclusion Criteria:

* Meets the age requirement and is in good health.

Exclusion Criteria:

* Have related vitamin D metabolic diseases (kidney failure, severe liver damage, hereditary 1α hydroxylase deficiency, etc.).
* Have an immune system disorder.
* Have a history of disabling cerebrovascular disease.
* Have a grade 1 or 2 relative with PD.
* Have severe dementia, depression, or serious mental illness.
* Failure to sign the informed consent form.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Th17 | Evaluation at the time of enrollment and intervention after three months.
  Detect the level of Th17 in peripheral blood.
Treg | Evaluation at the time of enrollment and intervention after three months.
  Detect the level of Treg in peripheral blood.
Vitamin D | Evaluation at the time of enrollment and intervention after three months
  Detect the level of Vitamin D in peripheral blood.

SECONDARY OUTCOMES:
UPDRS | Evaluation at the time of enrollment and intervention after three months
  Each item in the UPDRS (Unified Parkinson's Disease Rating Scale) is scored on a scale of 0 to 4, with 0 indicating normal and 4 indicating the most severe symptoms. The UPDRS can be divided into four subscales: the first subscale is used to assess the degree of mental activity, behavior, and emotional disorders in Parkinson's disease patients; the second subscale evaluates the patients' ability to perform activities of daily living; the third subscale, known as UPDRS-III, is the focus of the UPDRS scoring and assesses the motor function of PD patients, using 18 sub-items and a total of 132 points to describe the main motor symptoms of Parkinson's disease; the fourth subscale is used to evaluate treatment-related complications that occur during the course of PD treatment.
Berg balance scale | Evaluation at the time of enrollment and intervention after three months.
  This scale consists of 14 items, each scored from 0 to 4. The sum of these items gives a total score ranging from 0 to 56, with higher scores indicating better balance.
MMSE | Evaluation at the time of enrollment and intervention after three months
  This scale consists of 11 items, covering inquiries about orientation such as time and place, as well as assessments of memory, calculation ability, attention, recall ability, language skills, and visuospatial abilities. The language test further includes sub-tests for repetition ability, naming ability, command comprehension, reading ability, and writing ability. The total score for the MMSE is 30, and the entire test takes about 8-10 minutes to complete. A higher score indicates better cognitive function.
MoCA | Evaluation at the time of enrollment and intervention after three months
  It is an assessment tool used for rapid screening of cognitive dysfunction. It covers eight cognitive domains: visuospatial skills, executive function, memory, language, attention and concentration, calculation, abstract thinking, and orientation. The total score is 30, with a score of ≥26 considered normal.
SDS | Evaluation at the time of enrollment and intervention after three months
  This scale is an effective clinical tool for measuring subjective feelings of depression. It is a self-rating scale consisting of 20 items, each rated on a 4-point scale.
SAS | Evaluation at the time of enrollment and intervention after three months.
  This scale is a self-rating scale consisting of 20 items, each rated on a 4-point scale, used to assess the subjective feelings of patients with anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Hospital of Anhui Medical University, Suzhou, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li D, Ma X, Zhang W, Zhong P, Li M, Liu S. Impact of vitamin D3 supplementation on motor functionality and the immune response in Parkinson's disease patients with vitamin D deficiency. Sci Rep. 2025 Jul 11;15(1):25154. doi: 10.1038/s41598-025-10821-5. PMID 40646117